CLINICAL TRIAL: NCT07196449
Title: A Drug-drug Interaction Study to Evaluate the Effect of Rifampicin and Cyclosporine on the Pharmacokinetics of Methotrexate in Healthy Subjects
Brief Title: Drug-Drug Interaction of Rifampicin and Cyclosporine on Methotrexate Pharmacokinetics in Healthy Subjects
Acronym: MRCI
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Chung, Jae Yong, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MRCI
Record Dates: First submitted 2025-05-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Drug Drug Interaction (DDI)
Keywords: MRCI; Methotrexate; Rifampicin; Cyclosporine; DDI; Drug Drug Interaction
MeSH Terms: interventions — Methotrexate; Rifampin; Cyclosporine

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, 3-period, 6-sequence crossover Phase 1 clinical trial in healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): Sequence Group 1: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 1, Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 2, and Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 3 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration).
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine
- Group 2 (Experimental): Sequence Group 2: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 1, Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 2, and Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 3 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration).
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine
- Group 3 (Experimental): Sequence Group 3: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 1, Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 2 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration), and Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 3.
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine
- Group 4 (Experimental): Sequence Group 4: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 1, Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 2 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration), and Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 3.
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine
- Group 5 (Experimental): Sequence Group 5: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 1 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration), Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 2, and Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 3.
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine
- Group 6 (Experimental): Sequence Group 6: Two subjects assigned to this group will receive Methotrexate 2.5 mg + Cyclosporine 100 mg in Period 1 (1 subject with simultaneous administration, 1 subject with 1-hour staggered administration), Methotrexate 2.5 mg + Rifampicin 300 mg (single co-administration) in Period 2, and Methotrexate 2.5 mg + Rifampicin 150 mg (single co-administration) in Period 3.
  Interventions: Drug: Methotrexate; Drug: Rifampicin; Drug: Cyclosporine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate Tab. 2.5 mg (Korea United Pharm)
  Other Names: MTX
Drug: Rifampicin — Rifampin Cap. 150 mg (Yuhan Corporation)
  Other Names: RFP
Drug: Cyclosporine — Cypol-N Cap. 100 mg (Chong Kun Dang)
  Other Names: CsA

SUMMARY:
This study will evaluate how methotrexate is processed in the body when given with low doses of rifampicin or cyclosporine. These drugs may affect how methotrexate is absorbed and cleared, which could change its safety and effectiveness. Healthy volunteers will receive methotrexate with either rifampicin or cyclosporine, and blood samples will be collected to measure drug levels. The findings may help identify possible drug interactions and improve the safe use of methotrexate.

DETAILED DESCRIPTION:
Unexpected or unrecognized drug-drug interactions can reduce efficacy, cause toxicity, or even lead to fatal outcomes. Inhibition or induction of drug transporters involved in hepatic or renal uptake/efflux may alter drug exposure, affecting safety and efficacy. The FDA requires clinically significant interactions to be assessed prior to approval.

OATPs (primarily hepatic uptake) and BCRP (hepatic and renal efflux) share many substrates, but their combined inhibition has not been well studied in humans. Methotrexate, a substrate of both OATP and BCRP, is widely used at varying doses for cancer, psoriasis, and rheumatoid arthritis, often in combination with other drugs such as NSAIDs, which may result in interactions requiring close monitoring.

Rifampicin, an antibiotic, inhibits OATP1B1/1B3 in a dose-dependent manner, while cyclosporine, an immunosuppressant, inhibits OATP and BCRP. In our previous study (IRB No. B-2110-715-001), the investigators quantitatively demonstrated that rifampicin reduces 7-OH-methotrexate formation via OATP inhibition. However, dose-dependent inhibition by rifampicin and the impact of cyclosporine on methotrexate pharmacokinetics remain unclear.

This study aims to evaluate the pharmacokinetics of methotrexate following co-administration with low-dose rifampicin (150 or 300 mg) and cyclosporine in healthy volunteers. The investigators will also explore the role of methotrexate metabolites as potential biomarkers to assess OATP-mediated interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged between 19 and 45 years (inclusive) at the time of screening visit.
2. Body weight between 50.0 kg and 90.0 kg (inclusive) and a body mass index (BMI) between 18.0 and 30.0 kg/m² (inclusive) at the time of screening.

   ※ BMI (Body Mass Index) = weight (kg) / height² (m²)
3. Judged by the investigator to be suitable for participation in the study based on physical examination, clinical laboratory tests, and medical history.
4. Willingly provided written informed consent to participate after receiving and fully understanding a detailed explanation of the study prior to any screening procedures.

Exclusion Criteria:

1. Individuals with clinically significant hepatic (e.g., biliary obstruction), renal, neurologic, immunologic, gastrointestinal (e.g., irritable bowel syndrome, constipation), respiratory, endocrine disorders, or hematologic/oncologic, cardiovascular, or psychiatric disorders (e.g., mood disorders, obsessive-compulsive disorder), or relevant medical history.
2. History of clinically significant hypersensitivity to the investigational product, drugs in the same class, or other medications (e.g., aspirin, antibiotics) or food products.
3. History of gastrointestinal diseases (e.g., Crohn's disease, peptic ulcer) or surgeries that may affect drug absorption (except for simple appendectomy or hernia repair).
4. Known hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
5. Subjects meeting any of the following criteria at screening: AST(SGOT) or ALT(SGPT) > 1.5 × upper limit of normal (ULN); eGFR < 80 mL/min/1.73m² (calculated using CKD-EPI equation); QTc interval > 450 ms; Sitting blood pressure after ≥3 minutes of rest: systolic < 90 mmHg or > 150 mmHg, or diastolic < 50 mmHg or > 100 mmHg.
6. Total bilirubin > 1.8 mg/dL or serum potassium > 5.0 mmol/L (risk of hyperkalemia).
7. Positive results for HBsAg, anti-HCV, HIV (Ag/Ab), or RPR serologic tests.
8. History of drug abuse or positive results for drugs of abuse in urine screening.
9. Habitual alcohol consumption > 21 units/week (1 unit = 10 g pure alcohol), or unable to abstain from alcohol during the study.
10. Current smokers or those unable to abstain from smoking from 3 months prior to first dosing until the end of the study.
11. Use of enzyme or transporter inducers/inhibitors (e.g., barbiturates, statins, digoxin) within 3 months prior to the first dosing.
12. Unable to avoid St. John's Wort or grapefruit-containing products from 14 days before first dosing until study completion.
13. Habitual excessive caffeine intake (>5 units/day), or unable to abstain from caffeine or caffeine-containing products (e.g., coffee, tea, energy drinks) from 7 days before first dosing through the study.
14. Use of prescription drugs or herbal medicines within 2 weeks, or over-the-counter drugs, supplements, or vitamins within 10 days before first dosing (unless deemed acceptable by the investigator).
15. Participation in another clinical trial involving drug administration within 6 months prior to the first dosing day.
16. Whole blood donation within 2 months or component donation or transfusion within 1 month prior to the first dosing day.
17. Individuals with unusual dietary habits (e.g., strict vegetarians) or those unable to consume the provided meals entirely.
18. Individuals (male or female) of childbearing potential who are unable or unwilling to use acceptable contraception (e.g., surgical sterilization of self or partner, intrauterine device, hormonal contraception, diaphragm/condom with spermicide) during the study and for 2 weeks after the last dose of investigational product.
19. Any other condition that the investigator deems makes the subject unsuitable for study participation.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
MTX Cmax | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Peack plasma concentration (Cmax) of methotrexate
MTX AUClast | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Area under the concentration-time curve to last measurable concentration (AUClast) of methotrexate

SECONDARY OUTCOMES:
MTX AUCinf | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of Methotrexate
MTX Tmax | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Time to maximum plasma concentration (Tmax) of methotrexate
MTX t1/2 | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Terminal elimination half-life (t1/2) of methotrexate
MTX CL/F | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Apparent clearance (CL/F) of methotrexate
MTX Vz/F | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Apparent volume of distribution (Vz/F) of methotrexate
MTX fe | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Fraction of dose excreted unchanged in urine (fe) of methotrexate
MTX CLR | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Renal clearance (CLR) of methotrexate
7-OH MTX Cmax | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Maximum plasma concentration (Cmax) of 7-hydroxy methotrexate
7-OH MTX AUClast | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUClast) of 7-hydroxy methotrexate
7-OH MTX AUCinf | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of 7-hydroxy methotrexate
7-OH MTX Tmax | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Time to maximum plasma concentration (Tmax) of 7-hydroxy methotrexate
7-OH MTX t1/2 | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Terminal elimination half-life (t1/2) of 7-hydroxy methotrexate
7-OH MTX CL/F | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Apparent clearance (CL/F) of 7-hydroxy methotrexate
7-OH MTX Vz/F | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Apparent volume of distribution (Vz/F) of 7-hydroxy methotrexate
7-OH MTX fe | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Fraction of dose excreted unchanged in urine (fe) of 7-hydroxy methotrexate
7-OH MTX CLR | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Renal clearance (CLR) of 7-hydroxy methotrexate
7-OH MTX MR | pre-dose (0 hours), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, and 24 hours post-dose for each period (11 time points per period)
  Metabolic ratio (MR) of 7-hydroxy methotrexate

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Chung, Professor, Principal Investigator — Seoul National University Bundang Hospital, Department of Cliniacl Pharmacology
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea